CLINICAL TRIAL: NCT01809197
Title: Silicone Hydrogel Contact Lens Clinical and Comfort Benefits With a Multi-Purpose Disinfecting Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: M-12-056
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-06

CONDITIONS: Refractive Error; Myopia; Hyperopia; Astigmatism; Presbyopia
Keywords: Refractive error; Myopia; Hyperopia; Astigmatism; Presbyopia; Contact lenses; Contact lens solution; Comfort
MeSH Terms: conditions — Refractive Errors; Myopia; Hyperopia; Astigmatism; Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air Optix/OFPM (Experimental): Lotrafilcon B contact lenses (sphere, toric and multifocal), worn on a daily wear basis for 30 days, with OPTI-FREE MPDS lens care system
  Interventions: Device: Lotrafilcon B contact lenses; Device: OPTI-FREE PureMoist Multi-Purpose Disinfecting Solution (MPDS)
- Acuvue Oasys/Habitual MPS (Active Comparator): Senofilcon A contact lenses (sphere, toric and multifocal), worn on a daily wear basis for 30 days, with habitual MPS lens care system
  Interventions: Device: Senofilcon A contact lenses; Device: Habitual Multi-Purpose Solution (MPS)

INTERVENTIONS:
Device: Lotrafilcon B contact lenses — Silicone hydrogel contact lenses for near/far-sightedness, astigmatism, and/or presbyopia, replaced per manufacturer's instructions
  Other Names: AIR OPTIX® AQUA; AIR OPTIX® AQUA Multifocal; AIR OPTIX® for Astigmatism
  Arms: Air Optix/OFPM
Device: Senofilcon A contact lenses — Silicone hydrogel contact lenses for near/far-sightedness, astigmatism, and/or presbyopia, replaced per manufacturer's instructions
  Other Names: ACUVUE® OASYS® with HYDRACLEAR® PLUS; ACUVUE® OASYS® for ASTIGMATISM with HYDRACLEAR® PLUS; ACUVUE® OASYS® for PRESBYOPIA with HYDRACLEAR® PLUS
  Arms: Acuvue Oasys/Habitual MPS
Device: OPTI-FREE PureMoist Multi-Purpose Disinfecting Solution (MPDS) — Multi-purpose disinfecting solution for contact lens care, used per manufacturer's instructions
  Other Names: OPTI-FREE® PureMoist™
  Arms: Air Optix/OFPM
Device: Habitual Multi-Purpose Solution (MPS) — Multi-purpose solution for contact lens care according to subject's habitual brand, used per manufacturer's instructions
  Arms: Acuvue Oasys/Habitual MPS

SUMMARY:
The purpose of this study was to compare lens comfort on Day 30 for Air Optix® lenses cared for with OPTI-FREE® PureMoist® (OFPM) Multi Purpose Disinfecting Solution (MPDS) compared to Acuvue® Oasys® lenses cared for with habitual MPDS.

DETAILED DESCRIPTION:
Prior to the 30-day study period, subjects were fitted with study lenses in a masked manner and underwent a run-in period of 4-8 days to adjust to the randomized lenses.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent.
* Currently wearing weekly/monthly contact lenses on a daily wear basis, as specified in protocol.
* Willing to wear contact lenses on a daily wear basis for the duration of the study.
* Currently using a multi-purpose solution, as specified in protocol.
* Vision correctable to 20/30 (Snellen) or better in each eye at distance at Visit 1.
* Willing to follow the study procedures and visit schedule.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Currently wearing Air Optix, Acuvue Oasys, or Acuvue Advance brand of lenses.
* Currently using any Opti-Free brand of multi-purpose solution.
* Must wear contact lenses on an extended wear (overnight) basis during the study.
* Known sensitivity or intolerance to POLYQUAD® or ALDOX preserved lens care products.
* Monocular (only one eye with functional vision), fit with only one lens, or monovision modality of wear.
* Use of additional lens care products other than a multi-purpose solution within 7 days prior to Visit 1.
* Use of topical ocular over-the-counter (OTC) or prescribed topical ocular medications, with the exception of contact lens rewetting drops, within 7 days prior to Visit 1.
* Any abnormal ocular condition observed during the Visit 1 slit-lamp examination.
* Current or history of ocular infections (i.e., microbial keratitis, conjunctivitis) or severe inflammation (i.e., iritis, infiltrates) within the 6 months prior to Visit 1.
* Ocular surgery within the 12 months prior to Visit 1.
* Any systemic diseases at Visit 1 (including allergies, respiratory infections or colds) that affect the eye and could be exacerbated by use of contact lenses or contact lens solutions.
* Participation in any clinical study within 30 days of Visit 1.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Lemp, PhD, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 22 study sites located in the US.
Pre-assignment Details: Of the 387 enrolled, 15 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (372).
Period: Overall Study
Arm/Group | Air Optix/OFPM | Acuvue Oasys/Habitual MPS
Started | 187 | 185
Completed | 177 | 177
Not Completed | 10 | 8
Not completed — Lost to Follow-up | 4 | 2
Not completed — Adverse Event | 2 | 3
Not completed — Failed slit lamp exam | 1 | 0
Not completed — Non-Compliance | 1 | 1
Not completed — Decision Unrelated to an Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Product not available | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who were randomized and received study regimen (test or control). Note: 1 subject randomized to Acuvue Oasys was not dispensed with study lenses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Air Optix/OFPM | Acuvue Oasys/Habitual MPS | Total
Number analyzed (Participants) | 187 | 184 | 371
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (10.12) | 35.0 (11.14) | 33.7 (10.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 142 | 283
  Male | 46 | 42 | 88

OUTCOME MEASURES:

1. Primary Outcome: Likert Scale Questionnaire Item: "I Can Comfortably Wear my Lenses"
Description: Response of subject to a questionnaire item using a 5-point Likert scale, where 5=strongly agree and 1=strongly disagree.
Time Frame: Day 30; after 4 hours of lens wear
Population: This analysis population includes all subjects who were randomized and received study regimen (test or control) with a Day 30 response to this Likert item.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Air Optix/OFPM | Acuvue Oasys/Habitual MPS
Number analyzed (Participants) | 178 | 177
units on a scale | 4.2 (0.90) | 4.4 (0.66)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for duration of study (3 months). This analysis group includes all subjects who were randomized and received study regimen (test or control). Note: 1 subject randomized to Acuvue Oasys was not dispensed study lenses.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device. AE data were collected at each study visit.
Arm/Group | Air Optix/OFPM | Acuvue Oasys/Habitual MPS
Serious Adverse Events (participants affected / at risk) | 0/187 | 0/184
Other Adverse Events (participants affected / at risk) | 0/187 | 0/184

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.